CLINICAL TRIAL: NCT06393439
Title: The Effect of Virtual Hand Movements on Functional Tremor - a Pilot Study
Brief Title: Virtual Reality in Functional Movement Disorder
Acronym: VR-FMD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 36-115 ex 23/24
Record Dates: First submitted 2024-03-28; First posted 2024-05-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Functional Movement Disorder
Keywords: Tremor; Virtual Reality; Functional neurological disorder
MeSH Terms: conditions — Conversion Disorder; Tremor

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Functional Movement Disorder (Experimental)
  Interventions: Diagnostic Test: Virtual reality motor task
- Essential Tremor (Experimental)
  Interventions: Diagnostic Test: Virtual reality motor task
- Healthy Control (Experimental)
  Interventions: Diagnostic Test: Virtual reality motor task

INTERVENTIONS:
Diagnostic Test: Virtual reality motor task — After a short practice task, participants perform motor tasks in a virtual reality environment. Reaction time is used to assess task performance.

SUMMARY:
This study investigates the effect of virtual reality (VR) motor tasks on functional movement disorders.

DETAILED DESCRIPTION:
The investigators want to investigate how different display modes of virtual hands and the experimental manipulation of the visual representation of virtual hand movements affect (1) the performance of the hand movements (2) the tremor and (3) the subjective perception of the tremor.

There are three groups: Patients with functional tremor (FT), patients with essential tremor (ET) and healthy controls (HC). The study is carried out on one or two consecutive days. The first appointment is only made for patients with ET and FT and is used for the neurological examination and to assess the severity of the tremor. It takes place at the Outpatient Clinic for Movement Disorders at the University Clinic for Neurology in Graz and lasts a maximum of 30 minutes. The second appointment is at the Institute of Psychology at the University of Graz and requires the active participation of the respondent for 2.5 hours. Subjects are asked not to take any tremor-influencing medication on the day of the examination. HC will only attend the appointment at the Institute of Psychology.

First appointment:

* Clinical Global Impression - Severity Scale (CGI-S): 5-point Likert scale, clinicians assess the severity of the condition
* Patient Global Impression of Severity (PGI-S): 5-point Likert scale, patients assess the severity of the condition
* Fahn Tolosa Marin Tremor Rating Scale (FTM): assesses the tremor severity
* Simplified Version of the Functional Movement Disorders Rating Scale (S-FMDRS): assesses the severity of the functional tremor

Second appointment:

1. Questionnaires:

   * Simulator Sickness Questionnaire (SSQ): 4-point Likert scale, assesses nausea, oculomotor and visual disturbances, disorientation (2 timepoints: before and after VR tasks)
   * Edinburgh Handedness Inventory (EDI)
   * Questionnaire about sociodemographic data
   * Technology Usage Inventory (TUI): 7-point Likert scale, acceptance and use of technologies
   * Igroup Presence Questionnaire (IPQ): sense of presence in the VR
2. electroencephalogram (EEG) and surface-Electromyography (surface-EMG) of forearm muscles: run synchronously with the examinations
3. VR-tasks: all tasks are carried out in randomized order

   1. 3x3 matrix: individual fields light up in random order, participants are instructed to touch the fields in the given sequence as quickly as possible. 30 repetitions with a realistic VR-hand model and 30 repetitions with an abstract VR-hand model.
   2. 3x3 matrix: same task as (a) but after each repetition, participants must touch a field labeled "next" to continue the task. 30 repetitions.
   3. apple in a box: a virtual apple is to be placed in a virtual box using the hand with the weaker tremor, while the other hand is left resting on the table. 30 repetitions.
   4. apple in a box: same task as (c) but the resting hand is not visible. 30 repetitions.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of functional tremor (FT) or essential tremor (ET) or healthy control persons
* In patients with FT and ET: presence of a constant or intermittent tremor during the neurological examination

Exclusion Criteria:

* unclear tremor syndrome
* essential tremor plus (ET plus)
* conditions that interfere with EEG diagnostic (skin conditions, skin infections, wounds)
* reflex epilepsy
* cervical degeneration or chronic pain syndrome of the cervical spine
* severe somatic illness
* previous cerebral or head surgery
* implanted pacemaker or deep brain stimulation
* persons who are unable to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Task performance | 4 measurement points: abstract hand model without time pressure, abstract hand model with time pressure, realistic hand model without time pressure, realistic hand model with time pressure. Approximately 2.5 hours
  Reaction time in processing the VR task, measured in seconds

SECONDARY OUTCOMES:
Tremor duration | 5 measurement points: tasks a, b, c, d; Approximately 2.5 hours
  Duration of tremor during the motor task, expressed as % of movement time (only in FT and ET)
EEG | 10 measurement points: resting state before each motor task and during each motor task; Approximately 2.5 hours
  Changes in mu and beta event-related (de)synchronizations between motor tasks and right and left hemispheres
Subjective tremor severity on a visual analogue scale (VAS) | 6 measurement points: before and after each task; Approximately 2.5 hours
  Subjective tremor severity measured by a visual analogue scale (VAS) from 0 to 10 points, with higher scores indicating greater tremor severity
VR acceptance | 2 measurement points: before and after the VR examination, Approximately 2.5 hours
  Technology Usage Inventory (TUI): from 29 to 203 points, with higher scores indicating greater acceptance of technologies

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schwingenschuh, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Department of Neurology, Graz, Austria

IPD SHARING:
Plan to Share IPD: No